CLINICAL TRIAL: NCT00809263
Title: A Randomized, Double-blind, Placebo-controlled, Homeopathic Drug Proving Using a Crossover Design
Brief Title: Homeopathic Drug Provings
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Medicine Institute (Other)
Collaborators: Southwest College of Naturopathic Medicine (Other); Heel GmbH (Unknown)
Responsible Party: Steven Messer ND DHANP, Southwest College of Naturopathic Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: HDPSCNM2008
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: homeopathy; homeopathic drug proving; Document symptoms associated with administration of a homeopathic remedy.
MeSH Terms: interventions — Homeopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: homeopathic remedy — Homeopathic remedy 12C potency, 10 drops TID X 7 days

SUMMARY:
In a homeopathic drug proving a homeopathically prepared substance is administered to healthy volunteers in order to produce the symptoms specific to that substance and thereby reveal its inherent curative powers. During a homeopathic drug proving the goal is to provoke temporary symptoms (or "artificial illness") associated with the homeopathic medication. These symptoms are then arranged to form a symptom pattern or 'remedy picture' which is specific to that particular homeopathic substance and provides the basis for a better understanding of the possible effects of that homeopathic remedy in patients.

DETAILED DESCRIPTION:
The duration of these homeopathic drug provings are six week per subject (42 days). The central investigational tool of the homeopathic drug proving is the journal kept by each subject from DAY 1-35. The subject describes the symptoms they experience in their own words in the journal daily. During the 7 day run-in phase, the subject notes in their journal their current state of health, the daily rhythm of their life, and any other signs or symptoms that occur on a daily basis. This will also enhance familiarity with self-observation and the recording of signs and symptoms. After completion of this run-in phase an evaluation including journal check will occur on DAY 7. During the following 4 weeks (observation periods DAY 8-14, 22-28; wash-out period DAY 15-21 and 29 - 35) the subject documents all signs or symptoms that occur in his/her journal on a daily basis. During this period, subject interviews will take place on DAY 15, DAY 21. DAY 29 and DAY 36. During the 7 day follow up (post observation period, DAY 36-42) the subject will be contacted to check if any additional symptoms and/or adverse events occurred.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and < 75 years
* General state of good health
* Continuation of the usual habits and patterns of daily living
* Written informed consent obtained and willingness to comply with the requirements of the study

Exclusion Criteria:

* Any major life changes e.g. moving, getting married or divorced etc.
* Current or expected medical treatment or surgery during this homeopathic drug proving
* Surgery within the past four weeks prior to enrollment into the homeopathic drug proving
* Use of homeopathic medicines > 30 C or contraceptive pills in the month prior to enrollment into the homeopathic drug proving
* Alcohol or drug abuse
* Pregnancy or nursing (or anticipating pregnancy during this homeopathic drug proving)
* Incompetence, or inability of understanding the nature, meaning and consequences of the homeopathic drug proving or inadequate completion of the journal form DAY 1-7.
* Participation in another clinical trial at the same time or within the last 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms associated with the administration of homeopathic remedy to health subjects. | 6 weeks per subject

CONTACTS AND LOCATIONS:
Overall Officials: Steven Messer, ND, Principal Investigator — Southwest College of Naturopathic Medicine
Locations (1):
- Southwest College of Naturopathic Medicine, Tempe, Arizona, United States